CLINICAL TRIAL: NCT03821428
Title: Acupuncture for Relief of Gag Reflex in Patients Undergoing Transesophageal Echocardiography - a Randomized Placebo-controlled Trial
Brief Title: Acupuncture for Relief of Gag Reflex
Acronym: AcuGag
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BB 166/18
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Gagging During Transesophageal Echocardiography
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Needling of acupoints P6 and CV24 with indwelling permanent needles, withdrawn after TEE procedure
  Interventions: Procedure: Acupuncture
- Control (Placebo Comparator): Application of Placebo needles in the areas of P6 and CV24 acupoints
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Acupuncture — Needling of P6 and CV24 points
  Other Names: Verum acupuncture
  Arms: Acupuncture
Procedure: Placebo — Application of placebo acupuncture needles to the areas, where the acupoints are situated
  Other Names: Placebo acupuncture
  Arms: Control

SUMMARY:
The aim of the study is to test whether stimulation of acupuncture points CV24 and P6 is better than placebo acupuncture in treatment of gagging in patients undergoing elective transesophageal echocardiography (TEE)

DETAILED DESCRIPTION:
Patients undergoing elective transesophageal echocardiography (TEE) often report discomfort because of active gagging reflex, which sometimes preclude the performance of TEE and requires additional medication. According to existing literature, needling of acupoint CV24 effectively prevents gagging during dental procedures. We are going to use this phenomenon in patients scheduled to TEE in order to reduce discomfort during insertion of TEE probe and reduce the need for additional sedative medication. Within this investigation the patients will be randomly assigned to receive either verum acupuncture of CV24 and P6 acupoints or placebo procedure immediately before TEE examination. As outcome the incidence and intensity of gagging, total dose of additional sedative medication and hemodynamic parameters will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an American Society of Anesthesiologists physical status of I to III scheduled for elective ambulatory transesophageal echocardiography (TEE) without sedation
2. TEE time does not exceed 30 minutes
3. Patients without previous opioid and psychotropic medication
4. Patients aged between 30 and 65 years, able to use visual analogue scale 100 mm
5. Patients who have given written informed consent

Exclusion Criteria:

1. Current psychiatric disease
2. Local skin infection at the sites of acupuncture
3. Aged < 30 or > 65 years
4. TEE time more than 30 min
5. Patients who consumed opioid medication at least 6 months before surgery
6. Patients with the history of: i) psychiatric disease; ii) insulin-dependent diabetes mellitus; iii) radio- or chemotherapy; iv) peripheral polyneuropathy.
7. Patients who are unable to understand the consent form or to use visual analogue scale 100 mm

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-13 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of gagging during probe insertion | 10 minutes after TEE probe insertion
  Incidence of gagging during TEE probe insertion: yes=1; no=2

SECONDARY OUTCOMES:
Gagging score | 10 minutes after TEE probe insertion
  Gagging score on Verbal Rating Scale from 0 to 10, where 0=no discomfort from TEE probe; 10=maximal discomfort during TEE probe insertion
Rescue medication | 10 minutes after TEE probe insertion
  Use of midazolam as rescue medication, given as a summary dose of required midazolam from minimum 1 milligram to maximum 10 milligram

CONTACTS AND LOCATIONS:
Overall Officials: Taras Usichenko, Study Chair — University Medicine of Greifswald
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No